CLINICAL TRIAL: NCT01466608
Title: Lipid Lowering Effect, and Lipidomic Profiles by Genotype of OATP1B1 and BCRP After Administration of Rosuvastatin in Patients With Hyperlipidemia
Brief Title: Influence of OATP1B1 and BRCP Genotype on Rosuvastatin PK, PD and Lipidomics in Hyperlipidemic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Young Min Cho, Assistant professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUCPT11_Rosuvastatin_Pt
Record Dates: First submitted 2011-10-27; First posted 2011-11-08 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Hypercholesterolemia
Keywords: OATP1B1; Rosuvastatin; lipidomics; pharmacodynamics
MeSH Terms: conditions — Hypercholesterolemia | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rosuvastatin (Experimental): Rosuvastatin 20 mg will be administered once a day for 8 weeks (open-label, one-arm, single-sequence design)
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — Oral administration of rosuvastatin 20 mg once daily for 21 days.
  Other Names: Crestor Tablet 20 mg manufactured by Astrazeneca

SUMMARY:
The aim of this study is to investigate the pharmacokinetics, lipid lowering effect and lipidomic profiles of 8-weeks rosuvastatin treatment by OATP1B1 genotype in hyperlipidemia patients.

DETAILED DESCRIPTION:
Within 3 weeks prior to the first administration of study drug, volunteers who agreed the participation of this study by their written consent will undergo screening, including physical examination and clinical laboratory test etc, to evaluate whether they are eligible to participate in this study. Study drugs will be administered at about 9 A.M. in the morning of the first drug administration day, after blood collection for evaluation of pharmacokinetics, lipid profiles, metabolomics and urine collection for metabolomic and genetic analyses.

Subjects should take the investigational product by themselves every morning for 8 weeks. On the days of 2nd, 4th, 6 and 8th week, blood collection for evaluation of pharmacokinetics, lipid profiles, metabolomics and urine collection for metabolomics will be conducted by visiting the clinical trials center. On the days of 2nd, 4th and 6th week, the study drug will be taken after blood and urine collection.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 35 to 55 years at the time of screening
* Serum LDL cholesterol (LDL-C) level ≤130 mg/dL
* Must be reliable and willing to make themselves available during the study period
* Must be willing to give blood sample for genotyping

Exclusion Criteria:

* A subject with present clinical manifestation or past medical history of hepatic, renal, respiratory, neurologic, hematologic, oncologic, psychiatric, cardiovascular or endocrine disease, except hyperlipidemia and mild hypertension (SBP < 160 mmg, DBP <100 mmHg).
* Administration of lipid lowering agent within 2 weeks before the first study drug administration.
* A subject with a history of gastrointestinal disease or surgery (except simple appendectomy or repair of hernia), which could influence the absorption of the study drug.
* A subject with a history of drug abuse, or a positive urine drug screening test
* A subject who takes or should take any medication that can influence lipid lowering effects or metabolic profiles of the study drug during the study period. (Investigators judge the wash-out period of the previously used medication before the administration of the study drug.)
* A subject who has participated in any other clinical trial within 3 months before the study drug administration.
* A subject who is judged to be ineligible to participate in the study due to abnormal clinical laboratory results or other reasons by investigators.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2011-11; Primary Completion 2013-01 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Changes of serum lipid levels from baseline for 8 weeks | Day 1, Day 15, Day 29, Day 43, Day 57
  Changes of serum total cholesterol, LDL-cholesterol, HDL-cholesterol and triglyceride levels at fasting from baseline to Day 1, Day 15, Day 29, Day 43, Day 57

SECONDARY OUTCOMES:
Urinary and plasma levels of the lipid metabolites for 8 weeks | Day 1, Day 15, Day 29, Day 43, Day 57
  The levels of the lipid metabolites in the samples collected prior to daily rosuvastatin dose on Day 1, Day 15, Day 29, Day 43, Day57 using UPLS-TOF-MS.

CONTACTS AND LOCATIONS:
Overall Officials: Young Min Cho, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Clinical Trials Center, Seoul National University Hospital, Seoul, South Korea